CLINICAL TRIAL: NCT01225575
Title: Prospective, Randomised, Open Label, Multicentre Phase II Clinical Trial to Investigate the Efficacy and Safety of the Treatment of Large Cartilage Knee Defects(4-10 cm²) With 3 Diff. Doses of the ACT Product co.Don Chondrosphere®
Brief Title: Assessment of Efficacy and Safety of 3 Different Doses of co.Don Chondrosphere to Treat Large Cartilage Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: co.don AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cod 16HS14; 2009-016816-20 (EudraCT Number)
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Large Articular Cartilage Lesions of the Femoral; Condyle, Trochlea, Tibia or Retropatellar
Keywords: large cartilage defects; knee joint; femoral condyle, tibia, trochlear, retropatellar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- co.don chondrosphere®, 3-7 spheroids/cm2 (Active Comparator): co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes.
  The dose in group A is 3-7 spheroids/cm2 defect
  Interventions: Drug: co.don chondrosphere®
- co.don chondrosphere®,10-30spheroids/cm2 (Active Comparator): co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes.
  The dose in group B is 10-30 spheroids/cm2 defect
  Interventions: Drug: co.don chondrosphere®
- co.don chondrosphere®,40-70spheroids/cm2 (Active Comparator): co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes.
  The dose in group C is 40-70 Spheroids/cm2 defect
  Interventions: Drug: co.don chondrosphere®

INTERVENTIONS:
Drug: co.don chondrosphere® — co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes.
  The dose in group A is 3-7 spheroids/cm2 defect, in group B 10-30 spheroids/cm2 defect and in group C 40-70 spheroids/cm2 defect
  Other Names: ACT3D-CS

SUMMARY:
This is a prospective, randomised, open label, multicentre Phase II clinical trial to investigate the efficacy and safety of the treatment of large defects with 3 different doses of the autologous chondrocyte transplantation product co.don chondrosphere® (ACT3D-CS) in subjects with cartilage defects of the knee.

After screening visit patients were booked for arthroscopy and had their cells harvesting from healthy cartilage. After the arthroscopy the patients were randomised in one of the three dose-groups. The cells are cultivated for 8-10 weeks in vitro to develope 3-dimensional spheroids, that are transplanted in an open knee procedure (treatment surgery)into the defect. Patients of all dose groups subsequently followed the same rehabilitation program and had post-surgery visits. The 12-month-visit is defined as final assessment. Then patients have follow-up assessments up to 60 months.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age: between 18 and 50 years
2. Defect: isolated ICRS grade III or IV single defect on medial or lateral femoral condyle, trochlea, tibia and retropatellar defects, also OCD (in case of OCD: Bone grafting up to the level of the original bone lamella must be performed if bone loss exceeds 3 mm in depth)
3. Defect size: ≥ 4 to 10 cm2 after debridement to healthy cartilage; chondral lesions, including osteochondritis dissecans on femoral condyle, trochlea, tibia,retropatellar defects up to 6 mm in depth. Assessment with MRI at Screening and per estimation during arthroscopy prior to randomization
4. Nearly intact surrounding chondral structure around the defect as well as corresponding joint area
5. Informed consent signed by patient
6. Patient understands strict rehabilitation protocol and follow-up programme and is willing to follow it.
7. In case of pain, patient agrees to use only paracetamol mono- (max 4 g/day) or combination preparation and oral and/or topic NSAIDs during the trial and to discontinue the use of oral and/or topic NSAIDs and/or paracetamol combination preparation 1 week before each visit whereas the use of paracetamol mono-preparation (max 4 g/day) is allowed. However, in the morning of the visit day, no pain medication is allowed. However, in the morning of the visit day, no pain medication is allowed. Other pain medications are allowed during surgical operation and may be taken for a period not exceeding 4 weeks after surgery.

Exclusion Criteria:

1. Defects on both knees at the same time
2. Radiological signs of osteoarthritis
3. Any signs of knee instability
4. Valgus or varus malalignment (more than 5° over the mechanical axis)
5. Clinically relevant second cartilage lesion on the same knee
6. More than 50 % resection of a meniscus in the affected knee or incomplete meniscal rim
7. Rheumatoid arthritis, parainfectious or infectious arthritis, and condition after these diseases
8. Pregnancy and planned pregnancy (no MRI possible)
9. Obesity (Body Mass Index >30)
10. Uncontrolled diabetes mellitus
11. Serious illness
12. Poor general health as judged by physician
13. Participation in concurrent clinical trials or previous trials within 3 months of screening
14. Previous treatment with ACT in the affected knee
15. Microfracture performed less than 1 year before screening in the affected knee
16. Alcohol or drug (medication) abuse
17. Meniscal transplant in the affected knee
18. Meniscal suture (in the affected knee) three months prior to baseline
19. Mosaicplasty (Osteoarticular Transplant System, OATS) in the affected knee
20. Having received hyaluronic acid intra-articular injections in the affected knee within the last 3 months of baseline
21. Taking specific osteoarthritis drugs such as chondroitin sulfate, diacerein, n-glucosamine, piascledine, capsaicin within 2 weeks of baseline
22. Corticosteroid treatment by systemic or intra-articular route within the last month of baseline or intramuscular or oral corticosteroids within the last 2 weeks of baseline
23. Chronic use of anticoagulants
24. Any concomitant painful or disabling disease of the spine, hips or lower limbs that would interfere with evaluation of the afflicted knee
25. Any clinically significant or symptomatic vascular or neurological disorder of the lower extremities
26. Any evidence of the following diseases in the affected knee: septic arthritis,inflammatory joint disease, recurrent episodes of pseudogout, Paget's disease of bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders, collagen gene mutation
27. Current diagnosis of osteomyelitis, human immunodeficiency virus (HIV-1, 2) and/or hepatitis C (HCV) infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of overall KOOS | 12 months after transplantation
  Change of overall KOOS (Knee Injury and Osteoarthritis Outcome Score) from baseline (Day 0)to final assessment (FA)determined for each dosage group and between the dosage groups.

SECONDARY OUTCOMES:
Change of overall KOOS | 24, 36, 48, 60 months after transplantation
  Change of overall KOOS from baseline (Day 0) to 24,36, 48 and 60 months follow-up, FU) after transplantation determined for each dosage group and compared between the dosage groups
Change of the 5 subscores of the KOOS | 12, 24, 36 ,48, 60 months after transplantation
  Change of the 5 subscores of the KOOS (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec), knee related Quality of life (QoL)) determined for each dosage group and between the dosage groups
Assessment of MRIs by the MOCART-Score (MRI Score) | 12, 24, 36, 48 and 60 months after transplantation
  Assessment of MRIs by the MOCART-Score (MRI Score) at 12, 24, 36, 48 and 60 months after transplantation compared between the dosage groups
Assessment of cartilage repair using an Arthroscopy and take a biopsy | 12 months after transplantation
  Arthroscopy and biopsy at 12 months after transplantation, assessment of cartilage repair after ACT3D to be compared for each dosage group and between the dosage groups
Assessment of the histology from the biopsy by ICRS Visual Histological Assessment Score | 12 months after transplantation
  Assessment of the ICRS Visual Histological Assessment Score at final assessment (FA, 12 months) determined for each dosage group and compared between the dosage groups
Assessment of the histology from the biopsy by the Bern Score and additional histological scores | 12 months after transplantation
  Assessment of the histology from the biopsy by the Bern Score and additional histological assessment scores at final assessment (12 months) determined for each dosage group and compared between the dosage groups
Change of ICRS/IKDC | 12, 24, 36, 48 and 60 months after transplantation
  Change of ICRS/IKDC from baseline (Day 0) to 12, 24, 36, 48 and 60 months after transplantation determined for each dosage group and compared between the dosage groups
Assessment of change of modified Lysholm Score | 12, 24, 36, 48 and 60 months after transplantation
  Change of modified Lysholm Score from baseline (Day 0) to 12, 24, 36, 48 and 60 months after transplantation determined for each dosage group and compared between the dosage the groups
Days of absence from work (employment) and/or days of inability to follow usual activities | annual
  Days of absence from work (employment) and/or days of inability to follow usual activities during the last year or since the last visit, respectively, and time point when patient was back to work and/or to follow usual activities
Frequency and type of adverse events | 3,12, 24, 36, 48, 60 months after transplantation
  Frequency and type of adverse events
Measurement of blood pressure, pulse and laboratory parameters | 3, 6, 12, 24, 36, 48, 60 months after transplantation
  Measurement of the vital signs and physical examination, laboratory parameters at 3 and 12 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Fickert, Ph.D., Principal Investigator — Universitätsmedizin Mannheim
Locations (10):
- Germany (10):
  - Universitätsklinikum der Albert-Ludwig-Universität Freiburg, Department Othopädie und Traumatologie, Freiburg im Breisgau, Baden-Würrtemberg
  - ATOS Klinikum Heidelberg, Zentrum für Knie- und Fußchirurgie, Heidelberg, Baden-Würrtemberg
  - Gelenk-und Wirbelsäulenzentrum Steglitz, Berlin
  - DRK-Kliniken Westend, Berlin
  - St. Vinzenz-Hospital, Dinslaken
  - Orthopädische Klinik der Medizinischen Hochschule Hannover, Hanover
  - Lubinus Clinicum Kiel, Kiel
  - DRK Krankenhaus Luckenwalde, Luckenwalde
  - Orthopädisch-Unfallchirurgisches Zentrum, Mannheim
  - Orthopädiezentrum München Ost, München

REFERENCES:
- [Derived] Hoburg A, Niemeyer P, Laute V, Zinser W, John T, Becher C, Izadpanah K, Diehl P, Kolombe T, Fay J, Siebold R, Fickert S. Safety and Efficacy of Matrix-Associated Autologous Chondrocyte Implantation With Spheroids for Patellofemoral or Tibiofemoral Defects: A 5-Year Follow-up of a Phase 2, Dose-Confirmation Trial. Orthop J Sports Med. 2022 Jan 18;10(1):23259671211053380. doi: 10.1177/23259671211053380. eCollection 2022 Jan. PMID 35071653
- [Derived] Becher C, Laute V, Fickert S, Zinser W, Niemeyer P, John T, Diehl P, Kolombe T, Siebold R, Fay J. Safety of three different product doses in autologous chondrocyte implantation: results of a prospective, randomised, controlled trial. J Orthop Surg Res. 2017 May 12;12(1):71. doi: 10.1186/s13018-017-0570-7. PMID 28499391
- [Derived] Niemeyer P, Laute V, John T, Becher C, Diehl P, Kolombe T, Fay J, Siebold R, Niks M, Fickert S, Zinser W. The Effect of Cell Dose on the Early Magnetic Resonance Morphological Outcomes of Autologous Cell Implantation for Articular Cartilage Defects in the Knee: A Randomized Clinical Trial. Am J Sports Med. 2016 Aug;44(8):2005-14. doi: 10.1177/0363546516646092. Epub 2016 May 20. PMID 27206690